CLINICAL TRIAL: NCT00335699
Title: A 6-Week, Randomised, Open-Label, Parallel Group, Multi-Centre Study to Compare the Efficacy of Rosuvastatin 10mg With Atorvastatin 10mg in the Treatment of Non-Diabetic Metabolic Syndrome Subjects With Raised LDL-C
Brief Title: Korean Rosuvastatin Effectiveness Study in Nondiabetic Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3560L00053; KREST
Record Dates: First submitted 2006-06-09; First posted 2006-06-12 (Estimated); Last update posted 2007-12-17 (Estimated); Status verified 2007-12

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia with nondiabetic metabolic syndrome
MeSH Terms: conditions — Hypercholesterolemia | interventions — Rosuvastatin Calcium

INTERVENTIONS:
Drug: Rosuvastatin

SUMMARY:
The primary objective of this study is to compare the effect of rosuvastatin 10mg with atorvastatin 10mg in the percentage reduction of LDL-C in Subjects with metabolic syndrome after 6 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Metabolic syndrome patient; Presence of 3 or more of the following:

  * Abdominal obesity (waist circumference): men > 90cm(36 inch), women > 80cm(32 inch)
  * Triglycerides ≥ 150 mg/dL (1.70 mmol/L)
  * HDL-C: men < 40 mg/dL (1.04 mmol/L), women < 50 mg/dL (1.3 mmol/L)
  * BP ≥130/≥85 mmHg or subject receiving anti-hypertensive treatment
  * Fasting blood glucose 110 mg dL (6.11 mmol/L) - 125 mg/dL (6.94 mmol.L)
* Elevated LDL-C concentrations reported within 4 weeks of visit 1 as follows;

  * ≥ 130 mg/dL (3.36 mmol/L) to < 220 mg/dL (5.69 mmol/L) in statin naive subjects (subjects who have not taken any lipid-lowering therapy known to affect LDL-C in the 4 weeks prior to visit 1)
  * ≥ 100 mg/dL (2.59 mmol/L) to < 160 mg/dL (4.14 mmol/L) in subjects who have taken a lipid lowering drug(s) within 4 weeks of visit 1
* Triglyceride levels < 400 mg/dL (4.52 mmol/L)
* Women of childbearing potential should be using a medically acceptable form of chemical or mechanical contraception.

Exclusion Criteria:

* History of known diabetes mellitus
* Use of anti-hyperglycaemic medication.
* History of serious or hypersensitivity reactions to HMG-CoA reductase inhibitors, in particular history of myopathy.
* No CHD or CHD Risk Equivalents and 0-1 Risk factors and Framingham 10-Year risk is <10%.
* History of heterozygous or homozygous familial hypercholesterolaemia or known type III hyperlipoproteinaemia (familial dysbetalipoproteinaemia).
* Active arterial disease such as unstable angina pectoris, myocardial infarction, transient ischaemic attack (TIA), cerebrovascular accident (CVA), coronary artery bypass surgery (CABG) or angioplasty within 2 months prior to entry in the dietary lead in period
* Uncontrolled hypothyroidism defined as thyroid stimulating hormone (TSH) > 1.5 times the upper limit of normal (ULN) at Visit 2 or subjects whose thyroid replacement therapy was initiated within 3 months of entry into dietary lead-in phase.
* Current active liver disease (alanine aminotransferase [ALT] > 2 x ULN) or severe hepatic impairment.
* Unexplained serum CK >3 times ULN (e.g. not due to recent trauma, intramuscular injections, heavy exercise, etc).
* Serum creatinine > 176 umol/L (2.0 mg/dL)
* History of alcohol, or drug, abuse or both.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370
Dates: Start 2005-08; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to compare the effect of rosuvastatin 10mg with atorvastatin 10mg in the percentage reduction of LDL-C in Subjects with metabolic syndrome after 6 weeks of treatment.

SECONDARY OUTCOMES:
The secondary objectives of this study are to compare the effects of rosuvastatin 10mg with atorvastatin 10mg in subjects with metabolic syndrome, after 6weeks of treatment, on:
Bringing subjects to their established NCEP ATP III target goals for LDL-C
Bringing subjects to their non-HDL target goal(based on NCEP-ATP III criteria)
Modifying other lipids and lipid ratios
Modifying inflammatory markers
Glucose and insulin resistance
Safety

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Korea Medical Director, MD, Study Director — AstraZeneca
Locations (7):
- South Korea (7):
  - Research Site, Daegu
  - Research Site, Iksan
  - Research Site, Jeonju
  - Research Site, Jinju
  - Research Site, Kwangju
  - Research Site, Pusan
  - Research Site, Ulsan